CLINICAL TRIAL: NCT02663206
Title: Peroral Endoscopic Myotomy Versus Botulinum Toxin Injection in the Treatment of Medical Refractory Spastic Esophageal Disorders
Brief Title: Peroral Endoscopic Myotomy Versus Botulinum Toxin Injection in Spastic Esophageal Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Eligible candidate for recruitment was not found
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00049663
Record Dates: First submitted 2016-01-05; First posted 2016-01-26 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Achalasia; Esophageal Spasm, Diffuse; Esophageal Motility Disorders
Keywords: spastic esophageal disorders; achalasia; diffuse esophageal spasm; hypercontractile (jackhammer) esophagus; Botulinum toxin injection; peroral endoscopic myotomy
MeSH Terms: conditions — Esophageal Achalasia; Esophageal Spasm, Diffuse; Esophageal Motility Disorders | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin injection (Other): Drug/Device: Botulinum toxin injection; Endoscopic Botulinum toxin (BTX) injection at lower esophagus; Upper endoscopy with Botulinum toxin injection.
  The procedure will be performed as an outpatient basis by an endoscopist. Sedation can be in form of conscious sedation, monitored anesthesia care or general anesthesia. An upper endoscope will be inserted into the patient's mouth and advanced into lower esophagus. Botulinum toxin (Botox@) 100 units 8-10 (25 units/mL) will be injected in 1-ml portion in each of four quadrants about 1 cm above the Z-line (the LES region).
  * At 1 month follow-up, patients who do not response to the first botox injection (Eckardt score > 3) will receive the second botox injection.
  * At 3-month follow-up, POEM will be offered as a rescue therapy to both non-responders (Eckardt score > 3 at 3-month follow-up after the procedure) and relapsers (Eckardt score ≤ 3 at 3-month follow-up but becomes > 3 during the follow-up)
  Interventions: Procedure: Botulinum toxin injection
- peroral endoscopic myotomy (Other): Procedure/Surgery: peroral endoscopic myotomy.
  The procedure will be performed by an endoscopist (gastroenterologist or surgeon). General anesthesia will be started and upper endoscope will be inserted into the patient's mouth and advanced into the stomach. Endoscopic myotomy will be performed. Mucosal entry will then be closed using endoscopic clips or endoscopic suturing.
  All patients will recover from their procedures according to standard practice. They will remain nothing per oral (NPO) the night after the procedure and started on intravenous proton pump inhibitors. A gastrografin esophagram will be obtained the next day and if no evidence of leak, the diet will be advanced to a soft diet for two weeks. The patients will be evaluated by study coordinator/PI on a daily basis during their hospitalization.
  Interventions: Procedure: peroral endoscopic myotomy

INTERVENTIONS:
Procedure: peroral endoscopic myotomy — peroral endoscopic myotomy
  Arms: peroral endoscopic myotomy
Procedure: Botulinum toxin injection — endoscopic Botulinum toxin (BTX) injection at lower esophagus
  Arms: Botulinum toxin injection

SUMMARY:
To compare the efficacy of peroral endoscopic myotomy and Botulinum toxin injection in spastic esophageal disorders.

DETAILED DESCRIPTION:
Spastic disorders of the esophagus encompass hyperactive conditions of the esophagus due to either abnormal premature contractions or extreme vigor. In the current iteration of the Chicago classification, spastic esophageal disorders include spastic (type III) achalasia, diffuse esophageal spasm (DES), and hypercontractile (jackhammer) esophagus. Management of these spastic esophageal disorders is challenging and not clearly defined. Several medical therapies have been suggested and include acid suppression, nitrates, muscle relaxants, and visceral analgesics. For those who fail to response to medical therapy, the treatment options are limited.

Botulinum toxin (BTX) injection is an effective therapeutic option for spastic esophageal disorders, however many patients experience symptoms relapse with this treatment requiring repeated injections.

Heller myotomy is a surgical option for patients with esophageal spastic disorders. As compared to other types of achalasia, the response rate to surgical myotomy was lower in patient with spastic achalasia. The theoretical reason for this is that the disease involves not only the lower esophageal sphincter (LES) but also the esophageal body. Given data to suggest that surgical myotomy may be effective in treating patients with spastic esophageal disorders, peroral endoscopic myotomy (POEM), which is a less invasive treatment modality, has recently been studied for these difficult-to-treat patients. An initial study reported high success rate of POEM for severe spastic esophageal disorders. The response rate as defined by Eckardt score to ≤ 3 was 96% in spastic achalasia, 100% in DES and 70% in those with Jackhammer esophagus after a median follow-up of 234 days in a largest case series of medically refractory spastic esophageal disorders.

To date, the optimal treatment for patients with severe symptomatic esophageal spastic disorders who fail medical therapy is unclear. Here, investigators aim to compare POEM and BTX injection in a randomized design.

To compare the efficacy of peroral endoscopic myotomy and Botulinum toxin injection in spastic esophageal disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age 18 - 80 years old.
2. Spastic disorders of the esophagus include spastic (type III) achalasia, distal esophageal spasm (DES), and hypercontractile (jackhammer) esophagus via high resolution esophageal manometry (HRM) 2.

   * DES is characterized by normal esophagogastric junction relaxation (integrated relaxation pressure [IRP] <15 mm Hg) and ≥ 20% premature contractions.
   * Spastic achalasia is defined as impaired EGJ relaxation (IRP ≥15 mm Hg) associated with ≥ 20% premature contractions.
   * The diagnosis of jackhammer esophagus is defined as at least 1 swallow with a distal contractile integral (DCI) greater than 8000 mm Hg- s- cm.
3. At least 6 months of symptoms (chest pain, dysphagia, regurgitation and/or weight loss) with no adequate response or intolerance to medical therapy including nitrates and/or calcium channel blockers.
4. Overall symptoms score (Eckardt score) > 3
5. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Diagnosis of spastic esophageal disorder was not confirmed by HRM testing.
2. Previous surgery of the esophagus or stomach
3. Previous BTX injection at the esophagogastric junction (EGJ) or LES.
4. Active severe esophagitis
5. Large lower esophageal diverticula
6. Large > 3cm hiatal hernia
7. Megaesophagus (> 6 cm)
8. Sigmoid esophagus
9. Known gastroesophageal malignancy
10. Inability to tolerate sedated upper endoscopy due to cardiopulmonary instability, severe pulmonary disease or other contraindication to endoscopy
11. Cirrhosis with portal hypertension, varices, and/or ascites
12. Uncorrectable coagulopathy defined by prothrombin time < 50% of control; partial thromboplastin time (PTT) > 50 sec, or international normalized ratio (INR) > 1.5), on chronic anticoagulation, or platelet count <75,000.
13. Pregnant or breastfeeding women (all women of child-bearing age will undergo urine pregnancy testing)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Eckardt score | 3-month
  symptoms scores

SECONDARY OUTCOMES:
Eckardt score | 1-year
changes in individual symptom scores | 3 months and 12 months
  Each symptoms scores that are used to calculated Eckardt score
changes in esophageal manometry | 3 months
rate of complications | 3 months and 12 months
quality of life scores | 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A Khashab, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States